CLINICAL TRIAL: NCT01553968
Title: Effects of Acute Exercise on Acetylcarnitine Concentration in Endurance Trained and Untrained Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-2-069
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endurance Trained Subjects (Other)
  Interventions: Other: Cycling
- Untrained Subjects (Other)
  Interventions: Other: Cycling

INTERVENTIONS:
Other: Cycling — 30 minutes of cycling at 50% of predetermined maximal performance

SUMMARY:
It has been suggested that imbalance between TCA-cycle flux and β-oxidation may underlie insulin resistance, a predisposing factor for the development of type 2 diabetes mellitus. Acetylcarnitine concentration is suggested to be a marker of such imbalance. It is expected that when TCA-cycle capacity is high (a high oxidative capacity), less acetylcarnitine will accumulate, because of an improved balance between supply and demand of lipids.

The major research objective is to examine if acute exercise results in a more pronounced increase in acetylcarnitine concentration in sedentary subjects compared to endurance-trained subjects and if the exercise-induced increase in acetylcarnitine is restored more quickly in endurance-trained subjects when compared to sedentary subjects.

The investigators hypothesize that the increase in acetylcarnitine levels will be lower in trained subjects when compared to sedentary subjects, due to a better balance between lipid supply and utilization by the TCA-cycle. Furthermore it is expected that acetylcarnitine concentrations will be restored faster in these trained subjects, because of a tighter regulation of influx of fatty acids.

To test this hypothesis the investigators want to compare the acetylcarnitine response to exercise in a group of sedentary subjects and a group of endurance trained subjects. This response will be measured for 30 minutes after exercise with the use of 1H-MRS.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI 18-25 kg/m2)
* Healthy
* Stable dietary habits
* No use of medication
* VO2-max for trained subjects above 50 mL/min/kg
* VO2-max for untrained subjects below 40 mL/min/kg

Exclusion Criteria:

* Any medical condition requiring treatment and/or medication use OR diminishing exercise tolerance
* Alcohol consumption of more than 20 g per day (± 2 units)
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in another biomedical study within 1 month prior to the screening visit
* Contraindications for MRI scan:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker of defibrillator
  * Cochlear implant
  * Iron- containing corpora aliena in the eye or brain
  * Hearing aids and artificial (heart) valves which is contraindicated for MRS
* Subjects, who do not want to be informed about unexpected medical findings cannot participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Exercise-induced changes in acetylcarnitine concentrations and dynamics of acetylcarnitine restoration after exercise | During 30 minutes prior to the exercise and for 30 minutes after exercise
  Acetylcarnitine concentration measured with Proton Magnetic Resonance Spectroscopy (1H-MRS)

SECONDARY OUTCOMES:
Substrate oxidation | Measured during the 30 minutes of exercise
  Measured with indirect calorimetry
Blood plasma free fatty acids | At the start and at the end of 30 minutes of exercise
  Blood sample of 10 mL
Blood plasma triglycerides | At the start and at the end of 30 minutes of exercise
  Blood sample of 10 mL
Blood plasma glucose | At the start and at the end of 30 minutes of exercise
  Blood sample of 10 mL

CONTACTS AND LOCATIONS:
Overall Officials: Vera B. Schrauwen-Hinderling, PhD., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands